CLINICAL TRIAL: NCT01334385
Title: OEF/OIF Veterans' Experiences of Habituation to Painful Stimuli, Perceived Burdensomeness and Failed Belongingness
Brief Title: Operation Enduring Freedom/Operation Iraqi Freedom Veterans' Experiences of Habituation to Pain, Perceived Burdensomeness, and Failed Belongingness
Status: Completed | Type: Observational
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Collaborators: University of Colorado, Denver (Other); Portland State University (Other); University of Missouri, Kansas City (Other)
Responsible Party: Lisa A. Brenner, Ph.D., ABPP, VA VISN 19 MIRECC; University of Colorado Denver- School of Medicine
Other Study IDs: 06-1080
Record Dates: First submitted 2011-04-11; First posted 2011-04-13 (Estimated); Last update posted 2011-04-13 (Estimated); Status verified 2011-04

CONDITIONS: Suicide
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- OEF/OIF Veterans through VA ECHCS

SUMMARY:
Veterans possess significant risk factors for self-directed violence (SDV). For example, depressed Veterans are at a greater risk for SDV than the general population. Although depressed male Veterans die by suicide at a higher rate than do their female counterparts (Zivin et al., 2007), female Operation Enduring Freedom/Operation Iraqi Freedom (OEF/OIF) Veterans are at higher risk for depression than males (Seal et al., 2009). Joiner's (2005) theory states that suicidal individuals (a) perceive themselves to be unbearable burdens onto others; (b) view their efforts at establishing and maintaining social connections as having been thwarted or failed; and (c) have developed the ability to engage in SDV due to from increased habituation to pain. This two-part study uses semi-structured interviews in an effort to determine the extent to which Joiner's theory is applicable to OEF/OIF Veterans. Part I of this study, which has been completed, assessed the components of this theory among primarily male OEF/OIF Veterans. Part II of this study is assessing this theory's components among female OEF/OIF Veterans. Participants were recruited from the female OEF/OIF Veteran population receiving services through the Eastern Colorado Health Care System (ECHCS). Comparisons across the interview responses will be made to identify commonalities among the participants' experiences.

DETAILED DESCRIPTION:
This is a qualitative, interview-based study designed to determine the extent to which three theoretical constructs - habituation to painful stimuli, perceived burdensomeness, and failed belongingness - are relevant to female veterans who have returned from OEF/OIF deployments. Joiner (2005) has proposed that the combination of those three factors is necessary and sufficient for an individual to engage in self-harm behaviors. Part I of this study, which explored Joiner's model among primarily male Veterans, is complete. Part II of the study will be a replication of Part I, but will instead be exploring Joiner's model in a female veteran population. The intention is to conduct a series of studies leading up to a full test of Joiner's model in a veteran population. OEF/OIF female veterans will be interviewed in an effort to determine how they understand these constructs and the language they use in discussing them.

Parts I and II of this study are necessary to determine that the key constructs are pertinent to veterans' experiences in general. It is also essential to identify the language they use when talking about these constructs. This information may be used in future studies to design veteran-specific measures. Using language which is meaningful to the population being studied increases the validity of a new measure and is considered good psychometric procedure (DeVellis, 2003; Haynes, Richard, & Kubany, 1995). In addition, interviewing female veterans from the overall population of those receiving mental health services will increase the generalizability of future measures that are developed. Presuming Joiner's model is correct, participating in the interview may lead female veterans to spontaneously indicate that these factors could lead a person to think seriously about suicide. This possibility is despite the fact that the study will not be specifically targeting suicidal veterans or the fact that none of the questions ask about suicide or suicide-related behavior.

ELIGIBILITY:
Inclusion Criteria:

Part I:

1. OEF/OIF returned veteran
2. Age 18-55 years old
3. Active case in mental health services

Part II:

1. OEF/OIF returned veteran
2. Female
3. Age 18-55 years old

Exclusion Criteria:

1. Failure to correctly answer questions related to the informed consent process
2. Active psychosis diagnosed by primary clinician
3. Imminent suicidality

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Part I: Subjects were recruited from the population of over 250 OEF/OIF veterans with active cases in MHS within the Eastern Colorado Health Care System (ECHCS).
  Part II: Subjects were recruited from the population of over 250 OEF/OIF female veterans being cared for within the ECHCS.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2007-03; Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A Brenner, Ph.D., ABPP, Principal Investigator — VA Eastern Colorado Health Care System
Locations (1):
- VA Eastern Colorado Healthcare System, Denver, Colorado, United States